CLINICAL TRIAL: NCT06227338
Title: ICG-fluorescence Imaging for Intraoperative Breast Cancer Margins Evaluation: a Dose-timing Study
Acronym: BREASTIFLU-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJB-S2022-IFIBC01
Record Dates: First submitted 2023-09-21; First posted 2024-01-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Conservative surgery; Indocyanine Green
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Indocyanine green dye (Diagnostic Green) will be diluted with sterile water and a specific dose-arm (0.125 mg/kg, 0.25 mg/kg, 05 mg/kg, 1 mg/kg, and 2 mg/kg) will be administrated by slow intravenous injection by peripheral venous catheter:
  * at induction anaesthesia of the surgical procedure (0.125 mg/kg or 0.25mg/kg), or
  * in the hospital room 24 hours before the breast surgery (05 mg/kg, or 1 mg/kg, or 2 mg/kg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 0.125 mg/kg (Experimental): Patients who will be injected with 0.125 mg/kg Indocyanine green before their tumorectomy
  Interventions: Drug: Indocyanine green
- 0.25 mg/kg (Experimental): Patients who will be injected with 0.25 mg/kg Indocyanine green before their tumorectomy
  Interventions: Drug: Indocyanine green
- 0.5 mg/kg (Experimental): Patients who will be injected with 0.5 mg/kg Indocyanine green before their tumorectomy
  Interventions: Drug: Indocyanine green
- 1 mg/kg (Experimental): Patients who will be injected with 1 mg/kg Indocyanine green before their tumorectomy
  Interventions: Drug: Indocyanine green
- 2 mg/kg (Experimental): Patients who will be injected with 2 mg/kg Indocyanine green before their tumorectomy
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green dye (Diagnostic Green) will be diluted with sterile water and a specific dose-arm (0.125 mg/kg, 0.25 mg/kg, 05 mg/kg, 1 mg/kg, and 2 mg/kg) will be administrated by slow intravenous injection by peripheral venous catheter:
  * at induction anaesthesia of the surgical procedure (0.125 mg/kg or 0.25mg/kg), or
  * in the hospital room 24 hours before the breast surgery (05 mg/kg, or 1 mg/kg, or 2 mg/kg).

SUMMARY:
Designed in five-arm, single-center, prospective randomized, observational- interventional, open-label study which will evaluate patients with histological proven early-stage BC that will undergo planned BCS for their local treatment.

Two preoperatively times frames will be used for the administration of a total of 5 different indocyanine green (ICG) dose as a single dose-patient arm.

In the first time frame (intraoperative arms), the dose of, respectively 0.125 mg/kg and 0.25 mg/kg of ICG will be administered at induction anesthesia (at least 20 minutes before the BCS) in two subgroups.

In the second time frame, (preoperative arms), the dose of, respectively, 0.5 mg/kg, 1 mg/kg, and 2 mg/kg of ICG will be administered 24 h before surgery in 3 subgroups.

DETAILED DESCRIPTION:
The majority of breast cancer (BC) patients are diagnosed with an early-stage disease and are good candidates for breast-conserving surgery (BCS). Achieving adequate margins of excision is the most important component of BCS. Currently intra-operative margin assessment (IOMA) techniques used for margins evaluation in BC, either histological or imagistic is not accurate enough to predict the margins status of breast resected tumours and to guide surgery.

Fluorescence imaging (FI) using indocyanine green (ICG), a non-specific fluorophore, has also been reported to be a new, promising, non-invasive and relatively low cost technology to improving the accuracy of tumor detection during surgery in different clinical cancers, such as those of the liver, colon, ovaries, head and neck, lungs and breast. Furthermore ICG-FI can provide a real-time guidance during surgery and could establish corrects margins resection by improving the visual delineation between normal and tumoral tissues.

Only two clinical experience of ICG-FI for evaluating surgical margins in BC was reported. The group of Keating reported the first one, in a pilot study of 12 patients, after ICG intravenous (IV) injection (5mg/kg) they found that there was residual fluorescence in the tumoral bed in 6 out of 12 patients, but none of these patients had positive margins at definitive pathology. Recently, the investigators have reported the utility of ICG-FI after intraoperative ICG IV injection of 0.25 mg/kg for intraoperative breast surgical margin assessment during BCS. In a study of 35 BC patients, the investigators observed that the sensitivity (Se), specificity (Sp), and negative predictive value (NPV), of ICG-FI to predict margin involvement on the breast operative specimens were 100%, 60% and 100% respectively. Several important technical points exist in the experimental and clinical use of ICG-FI. There is a great variability of the published data regarding the baseline characteristics of the ICG use, like dosage and timing of administration (perioperative vs delayed). Furthermore, the fluorescence imaging system is usually different.

In this study, the investigators would like to emphasize and to get more precision about the optimal ICG doses and timing, which could increase the diagnostic accuracy of intraoperative ICG-FI for resection margins assessment during BCS, after intravenously ICG administration.

ELIGIBILITY:
Inclusion Criteria:

1. female;
2. age of ≥18 years;
3. histological diagnosis of ductal invasive breast cancer;
4. a primary early-stage invasive breast cancer (cT1 and/or cT2, assessed clinically and/or radiologically), without prior BC surgery of the actually affected breast;
5. ECOG Performance Status (PS) 0 or 1;
6. signed informed consent form (ICF) obtained prior to any study related procedure.

Exclusion Criteria:

1. advanced invasive breast cancer (cT3 and/or cT4);
2. in situ breast cancer disease;
3. lobular invasive breast cancer (at histology);
4. invasive breast cancer treated by neoadjuvant chemotherapy and/or endocrine therapy;
5. prior history of invasive or breast cancer of the actually affected breast in the past;
6. history of allergy or hypersensitivity to investigational product (active substance or ingredients);
7. history of allergy to iodine or to shellfish;
8. have apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal, or disseminated autonomy of the thyroid gland;
9. documented coronary disease
10. advanced renal insufficiency (serum creatinine >1.5 mg/dL);
11. chronic liver disease with the Child-Pugh class B or C ;
12. concurrent medication which reduces or increases the elimination of indocyanine green dye (ie, anticonvulsants, haloperidol, and heparin) during the 2 weeks before the expected operation;
13. pregnant or lactating women;
14. inability to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ICG-FI technique for the detection of positive (involved) surgical margins at the patient level | 2 years
  The sensitivity (Se), specificity (Sp), negative predictive value (NPV), false negative rate (FNR), FPR of the ICG-FI technique will be computed at the patient level

SECONDARY OUTCOMES:
Comparison of ICG-FI technique accuracy at different doses and timing | 2 years
  The sensitivity (Se), specificity (Sp), negative predictive value (NPV), false negative rate (FNR), FPR of the ICG-FI technique will be computed
Characterization of the breast tumor fluorescence (tumor-to- background fluorescence ratio) | 2 years
  Characterization of the appearance and intensity of fluorescence at the level of tumor cells
Evaluation of fluorescence intensity of axillary lymph nodes | 2 years
  The distribution of fluorescence intensity will be calculated depending on the type of axillary lymph node (LN) : sentinel vs other and respectively metastatic LN vs healthy LN)

CONTACTS AND LOCATIONS:
Overall Officials: Florin Pop, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium